CLINICAL TRIAL: NCT05462678
Title: Strategies and Techniques for the Rehabilitation of Memory Deficits in Patients With Multiple Sclerosis
Brief Title: Memory Rehabilitation Strategies in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE/PROG.698
Record Dates: First submitted 2022-07-04; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Multiple Sclerosis
Keywords: Cognitive Rehabilitation; Motor Rehabilitation; Cognitive Impairment
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Rehabilitation (Experimental): the first group carried out a training of CR by three memory modules of the Rehacom program (http://www.emsmedical.net).
  Interventions: Behavioral: Cognitive Rehabilitation
- Combined Training (Experimental): the second group followed a mixed training program with the use of the version of the verbal memory module of the Rehacom program combined with the MR training.
  Interventions: Behavioral: Combined Rehabilitation
- Motor Rehabilitation (Experimental): the third group carried out a traditional MR training.
  Interventions: Behavioral: Motor Rehabilitation

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation — Each patient performed two weekly sessions of 45 minutes each, for 12 weeks
  Arms: Cognitive Rehabilitation
Behavioral: Combined Rehabilitation — Each patient performed one session per week (45 minutes) of CR and one session per week of traditional MR training for 12 weeks.
  Arms: Combined Training
Behavioral: Motor Rehabilitation — Each patient performed two weekly sessions45 minutes each, for a total of 12 weeks.
  Arms: Motor Rehabilitation

SUMMARY:
The clinical characteristics of MS are extremely variable from one patient to another. In about 60% of cases, motor disabilities are associated with cognitive deficits. The present study aims to compare three forms of cognitive / motor rehabilitation in three groups of patients with MS: rehabilitation of verbal memory with the Rehacom program; combined rehabilitation, associating a motor rehabilitation path with the Rehacom program; only motor rehabilitation course. Aims of the study will be: to verify whether the combined cognitive / motor rehabilitation can induce a significantly greater improvement in the memory performance of patients with MS compared to rehabilitation alone; check whether any improvement is objectively verifiable by patients and the impact it may have on patients' quality of life; monitor these effects after 6 months.

For these purposes, three homogeneous groups of 20 patients each will be enrolled, diagnosed with MS according to Mc Donald's criteria revisited by Polman (2011). The study will be divided into an initial clinical, cognitive, emotional, quality of life and functional self-perception (T0) assessment. Subsequently, the patients assigned to the three conditions will be provided with the pre-established rehabilitation treatments for a total duration of 12 weeks; at the end, each patient will undergo an overall re-evaluation (T1). Finally, a further overall reassessment will be carried out after 6 months, aimed at follow-up monitoring (T2).

Statistical analyzes will be of two types:

Within Group (aimed at assessing any improvement in the cognitive performance of each group of patients by comparing the assessments at T0 with those at T1 and T2); Between Group (aimed at comparing the results obtained by each group with those of the other 2 groups at T0, T1, and T2).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS defined according to McDonald's diagnostic criteria revised in 2011.
* RRMS or SPMS phenotype.
* Language Italian mother tongue.
* EDSS score <6.0

Exclusion Criteria:

* Neurological or psychiatric pathologies other than MS that can interfere with cognitive functioning
* Clinical relapses in the three months prior to enrollment
* Severe mental illness
* Psychiatric disorders severe enough to interfere with cognitive functioning
* Medications Steroid therapy in the 3 months prior to enrollment
* Motor limitations Upper limb dysfunction (paralysis or tremor) that does not allow to hold the PC mouse
* Sensory limitations Visual acuity impaired enough to not allow reading of the instructions to the various tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Pre- and Post treatment and long term cognitive efficiency | 9-months
  The primary outcome of this study is the scores on the cognitive tasks (Minimal Assessment of Cognitive Functioning in Multiple Sclerosis -MACFIMS). For MACFIMS score ranges from 1 to 3 with higher scores corresponding to higher cognitive impairment.

SECONDARY OUTCOMES:
Pre- and Post-treatment and long term motor efficiency | 9-months
  The secondary outcome of this study is the scores on the gait and balance efficiency scales (Tinetti Scale -TS); For TS the score ranges from 0 to 28 with higher scores corresponding to higher efficiency.

OTHER OUTCOMES:
Pre- and Post-treatment and long term disability and overall quality of life | 9-months
  Tertiary outcome is the scores on the self-perceived quality of life assessed with World Health Organization Disability Assessment Schedule- WHO-DAS 2. For WHO-DAS 2 total score ranges from 0 to 100, with lower scores indicate lower levels of disability e better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Nocentini, MD, Study Director — I.R.C.C.S. "Santa Lucia" Foundation
Locations (2):
- Italy (2):
  - Santa Lucia Foundation I.R.C.C.S., Roma, Rm
  - I.R.C.C.S. "Santa Lucia" Foundation, Rome

REFERENCES:
- [Derived] Argento O, Piacentini C, Bossa M, Caltagirone C, Santamato A, Saraceni V, Nocentini U. Motor, cognitive, and combined rehabilitation approaches on MS patients' cognitive impairment. Neurol Sci. 2023 Mar;44(3):1109-1118. doi: 10.1007/s10072-022-06552-4. Epub 2022 Dec 21. PMID 36542204